CLINICAL TRIAL: NCT00282256
Title: A Phase 2, Open-Label, Multi-center Study to Assess the Pharmacokinetics, Long-Term Safety and Tolerability of Tacrolimus in Stable Pediatric Liver Transplant Patients Converted From a Prograf® Based Immunosuppression Regimen to a Modified Release (MR) Tacrolimus Based Immunosuppression Regimen
Brief Title: A Study of a Modified-Release Tacrolimus Based Immunosuppression Regimen in Stable Pediatric Liver Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 03-0-160
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-08

CONDITIONS: Liver Transplantation
Keywords: Child; Pharmacokinetics; Immunosuppression Drugs; Hepatic transplant; Liver Transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus MR (Experimental): Participants continued to receive their stable twice daily dose of tacrolimus twice daily on Day 1 through Day 7 and on Day 8 were converted to tacrolimus modified release (MR) once-daily in the morning for 7 days on a 1:1 (mg:mg) basis for their total daily dose. Patients who completed the 2-week pharmacokinetic treatment period were eligible to continue receiving tacrolimus MR as part of the extension treatment period of the study. The extended treatment period began on Day 15 and consisted of a single dose of tacrolimus MR once every morning through the end of the study.
  Interventions: Drug: tacrolimus modified release (MR); Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus modified release (MR) — Oral
  Other Names: Advagraf,; FK506E,; MR4,; FKMR,; Astagraf XL
Drug: tacrolimus — Oral
  Other Names: Prograf,; FK506

SUMMARY:
A study to assess the pharmacokinetics, safety and effectiveness of tacrolimus in stable pediatric liver transplant patients converted from a Prograf® based immunosuppression regimen to a modified release tacrolimus based immunosuppression regimen.

DETAILED DESCRIPTION:
A 1 arm study to assess the pharmacokinetics, and long-term safety and effectiveness of a modified release tacrolimus based immunosuppression regimen in stable pediatric liver transplant patients converted from a Prograf® based immunosuppression regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently receiving Prograf® based immunosuppressive therapy for liver transplantation.
* Patient has stable whole blood trough level concentrations of Prograf® and is clinically stable

Exclusion Criteria:

* Patient has previously received an organ transplant other than a liver
* Patient is currently receiving sirolimus immunosuppression therapy.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2004-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (5):
- United States (5):
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - New Orleans, Louisiana
  - New York, New York
  - Madison, Wisconsin

REFERENCES:
- [Background] Heffron TG, Pescovitz MD, Florman S, Kalayoglu M, Emre S, Smallwood G, Wisemandle K, Anania C, Dhadda S, Sawamoto T, Keirns J, Fitzsimmons W, First MR. Once-daily tacrolimus extended-release formulation: 1-year post-conversion in stable pediatric liver transplant recipients. Am J Transplant. 2007 Jun;7(6):1609-15. doi: 10.1111/j.1600-6143.2007.01803.x. PMID 17511684

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Stable liver transplant recipients aged 12 years or younger receiving tacrolimus based immunosuppression regimen.
Pre-assignment Details: Pharmacokinetic (PK) treatment period was 14 days. Participants who completed the PK period were eligible to continue receiving tacrolimus MR in the extended treatment period, from Day 15 through Month 54.
Period: Pharmacokinetic Treatment Period
Arm/Group | Tacrolimus MR
Started | 19
Received Tacrolimus | 19
Received Tacrolimus MR | 18
Completed | 18
Not Completed | 1
Not completed — Poor venous access | 1
Period: Extension Treatment Period
Arm/Group | Tacrolimus MR
Started | 18
Completed | 16
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: The pharmacokinetic evaluable set was defined as all patients who completed both pharmacokinetic profiles: one for tacrolimus, and one for tacrolimus MR.
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 8.6 (2.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5
Reason for End Stage Liver Disease [Number; unit: participants]
  Biliary Atresia | 5
  Acute Fulminant (Hepatic) Failure | 2
  Fulminant Hepatitis | 2
  Tyrosinemia | 2
  Unknown | 1
  Other | 6
Type of Current Transplant [Number; unit: participants]
  Whole Cadaver | 10
  Split Cadaver | 4
  Living Donor | 4
Re-transplant [Number; unit: participants]
  No | 16
  Yes | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 Hours (AUC0-24) for Tacrolimus
Description: The area under the concentration-time curve was calculated from whole blood tacrolimus concentrations for both tacrolimus and tacrolimus MR at steady state using the linear trapezoidal rule. The AUC0-24 for tacrolimus was calculated as the sum of the AUC0-12 and AUC 12-24 for the morning and afternoon doses.
Time Frame: For tacrolimus, Day 7 at 0 (pre-dose), 0.5, 1, 2, 3, 6, 8, 12 (pre-dose), 13, 14, 15, 18, 20, and 24 hours. For tacrolimus MR, Day 14 at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 15, 18, 20, and 24 hours post-dose.
Population: The pharmacokinetic evaluable set was defined as all patients who completed both pharmacokinetic profiles: one for tacrolimus, and one for tacrolimus MR. A complete pharmacokinetic profile was considered to be a profile that was adequate to determine AUC0-24, Cmax, and Cmin.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 18
ng*hr/mL
  Day 7: Tacrolimus | 198.2 (99.2)
  Day 14: Tacrolimus MR | 193.0 (78.0)
Statistical Analysis 1: Comparison: Tacrolimus MR; The method of analysis of variance was used for the comparisons of AUC0-24. Exposure at steady state was used for tacrolimus (defined as Day 7) and for tacrolimus MR (defined as Day 14). The natural log (ln) was used to transform AUC0-24 prior to analysis and the results were transformed back to the original scale for the presentation of results; Test type: Non-Inferiority or Equivalence — If the 90% CI for AUC0-24 was found to lie entirely within the 80% to 125% range, then the exposure between the two formulations was considered to be equivalent; Ratio of means = 100.9, 90% CI 2-sided [90.8 to 112.1] — Tacrolimus/tacrolimus MR ratio of natural log transformed means expressed as a percent

2. Secondary Outcome: Maximum Observed Concentration of Tacrolimus (Cmax)
Description: The maximum concentration was calculated from whole blood tacrolimus concentrations for both the tacrolimus and tacrolimus MR at steady state, without interpolation.
Time Frame: as for outcome 1
Population: Pharmacokinetic evaluable set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 18
ng/mL
  Day 7: Tacrolimus | 20.7 (13.3)
  Day 14: Tacrolimus MR | 15.2 (5.7)

3. Primary Outcome: Minimum Observed Concentration of Tacrolimus (Cmin)
Description: The trough (minimum) concentration of tacrolimus determined from the tacrolimus whole blood concentration value at the 12 hour post-dose concentration based on the evening dose (i.e., the 8 am concentration) for tacrolimus and the 24-hour time point post-dose for tacrolimus MR, prior to receiving the next dose.
Time Frame: Day 7 at 12 hours post-dose (tacrolimus) and Day 14 at 24 hours post-dose (tacrolimus MR).
Population: Pharmacokinetic evaluable set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 18
ng/mL
  Day 7: Tacrolimus | 5.9 (2.9)
  Day 14: Tacrolimus MR | 5.3 (2.6)
Statistical Analysis 1: Comparison: Tacrolimus MR; The method of analysis of variance was used for the comparisons of Cmin. Exposure at steady state was used for tacrolimus (defined as Day 7) and for tacrolimus MR (defined as Day 14). The natural log (ln) was used to transform Cmin prior to analysis and the results were transformed back to the original scale for the presentation of results; Test type: Non-Inferiority or Equivalence — If the 90% CI for Cmin was found to lie entirely within the 80% to 125% range, then the exposure between the two formulations was considered to be equivalent; Ratio of means = 91.8, 90% CI 2-sided [82.6 to 102.2] — Tacrolimus/tacrolimus MR ratio of natural log transformed means expressed as a percent

4. Primary Outcome: Patient Survival
Description: Patient survival was defined as any participant known to be alive at the end of the study.
Time Frame: From enrollment until the end of study (up to 54 months).
Population: The Modified Full Analysis Set included all patients who took at least 1 dose of tacrolimus MR formulation during the extended treatment period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 18
percentage of participants | 94.44 [83.86 to 100.00]

5. Primary Outcome: Graft Survival
Description: Graft survival was defined as any participant who did not meet the definition of graft loss, where graft loss was defined as graft failure (re-transplant) or participant death.
Time Frame: From enrollment until the end of study (up to 54 months).
Population: Modified full analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 18
percentage of participants | 94.44 [83.86 to 100.00]

6. Secondary Outcome: Time to Maximum Observed Concentration of Tacrolimus (Tmax)
Description: Time to reach the first observed maximum concentration of tacrolimus was calculated from whole blood tacrolimus concentrations for both tacrolimus and tacrolimus MR at steady state, without interpolation.
Time Frame: as for outcome 1
Population: Pharmacokinetic evaluable set.
Measure: Median (Full Range); unit: hours
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 18
hours
  Day 7: Tacrolimus | 1.0 [0.5 to 19.7]
  Day 14: Tacrolimus MR | 2.0 [0.9 to 6.0]

7. Secondary Outcome: Percentage of Participants With Biopsy-confirmed Acute Rejection
Description: Biopsy-confirmed acute rejection (BCAR) is defined as an episode of acute liver allograft rejection that was confirmed by biopsy results and was Banff grade ≥ I. Biopsies were graded by the pathologist at the clinical site according to the 1997 Banff criteria for grading of acute liver allograft rejection: Indeterminate: Portal inflammatory infiltrate that fails to meet the criteria for diagnosis of acute rejection; Grade I (Mild): Rejection infiltrate in a minority of the triads that is generally mild and confined within the portal spaces; Grade II (Moderate): Rejection infiltrate, expanding to most or all of the triads; Grade III (Severe): Rejection infiltrate, expanding to most or all of the triads, with spillover into periportal areas and moderate to severe perivenular inflammation that extends into the hepatic parenchyma and is associated with perivenular hepatocyte. necrosis
Time Frame: From enrollment until the end of study (up to 54 months).
Population: Modified full analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 18
percentage of participants | 16.67

8. Secondary Outcome: Time to Event for Patient Non-survival
Description: For participants who died on study, the median number of days from first dose of study drug to death due to any cause.
Time Frame: From enrollment until the end of study (up to 54 months).
Population: Participants in the modified full analysis set who died on study.
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 1
days | 1204.00 [1204.0 to 1204.0]

9. Secondary Outcome: Time to Event for Graft Non-survival
Description: For participants with graft loss, the median number of days from the first dose of study drug to graft loss. Graft loss was defined as graft failure (re-transplant) or participant death.
Time Frame: From enrollment until the end of study (up to 54 months).
Population: Participants in the modified full analysis set with graft loss.
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 1
days | 1203.00 [1203.0 to 1203.0]

10. Secondary Outcome: Time to First Biopsy-confirmed Acute Rejection
Description: For participants with a biopsy-confirmed acute rejection (BCAR), the median number of days from the first dose of study drug to the date of biopsy confirmation. BCAR is defined as an episode of acute liver allograft rejection that was confirmed by biopsy results and was Banff grade ≥ I. Biopsies were graded by the clinical site pathologist according to the 1997 Banff criteria for grading acute liver allograft rejection: Indeterminate: Portal inflammatory infiltrate that fails to meet the criteria for diagnosis of acute rejection; Grade I: Rejection infiltrate in a minority of the triads that is generally mild and confined within the portal spaces; Grade II: Rejection infiltrate, expanding to most or all of the triads; Grade III: Rejection infiltrate, expanding to most or all of the triads, with spillover into periportal areas and moderate to severe perivenular inflammation that extends into the hepatic parenchyma and is associated with perivenular hepatocyte necrosis.
Time Frame: From enrollment until the end of study (up to 54 months).
Population: Participants in the modified full analysis set with a biopsy-confirmed acute rejection.
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 3
days | 748.00 [729.0 to 773.0]

11. Secondary Outcome: Grade of Biopsy-confirmed Acute Rejection Episodes
Description: Biopsy-confirmed acute rejection (BCAR) is defined as an episode of acute liver allograft rejection that was confirmed by biopsy results and was Banff grade ≥ I. Biopsies were graded by the clinical site pathologist according to the 1997 Banff criteria for grading of acute liver allograft rejection: Indeterminate: Portal inflammatory infiltrate that fails to meet the criteria for diagnosis of acute rejection; Grade I (Mild): Rejection infiltrate in a minority of the triads that is generally mild and confined within the portal spaces; Grade II (Moderate): Rejection infiltrate, expanding to most or all of the triads; Grade III (Severe): Rejection infiltrate, expanding to most or all of the triads, with spillover into periportal areas and moderate to severe perivenular inflammation that extends into the hepatic parenchyma and is associated with perivenular hepatocyte necrosis. For participants with more than one biopsy-confirmed acute rejection episode, the worst case grade is reported.
Time Frame: From enrollment until the end of study (up to 54 months).
Population: Participants in the modified full analysis set with a biopsy-confirmed acute rejection.
Measure: Number; unit: participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 3
participants
  Grade I | 2
  Grade II | 1
  Grade III | 0

12. Secondary Outcome: Number of Participants Receiving Anti-lymphocyte Antibody Therapy for Acute Rejection
Description: Steroid-resistant rejection episodes were treated with anti-lymphocyte antibodies. If a participant had a histologically proven Banff Grade II or III rejection, they could be initiated on anti-lymphocyte antibody treatment per institutional practice.
Time Frame: From enrollment until the end of study (up to 54 months).
Population: Modified full analysis set.
Measure: Number; unit: participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 18
participants | 0

13. Secondary Outcome: Number of Participants With Multiple Rejection Episodes
Description: This analysis includes rejection episodes that were either confirmed by biopsy by the clinical site pathologist or were clinically treated.
Time Frame: From enrollment until the end of study (up to 54 months).
Population: Modified full analysis set.
Measure: Number; unit: participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 18
participants | 1

14. Secondary Outcome: Number of Participants With Clinically Treated Acute Rejection Episodes
Description: A clinically treated acute rejection episode was any biopsy-confirmed or suspected rejection episode that was treated with immunosuppressive therapy.
Time Frame: From enrollment until the end of study (up to 54 months).
Population: Modified full analysis set.
Measure: Number; unit: participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 18
participants | 3

15. Secondary Outcome: Number of Participants With Chronic Rejection
Description: Due to the low number of participants with biopsy-confirmed acute rejection episodes, chronic rejection was not analyzed.
Time Frame: From enrollment until the end of study (up to 54 months).
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 0

16. Secondary Outcome: Number of Participants With Treatment Failure
Description: Treatment failure was defined as discontinuation of study drug for any reason. Due to discontinuation of the study by the sponsor, treatment failure was not analyzed.
Time Frame: From enrollment until the end of study (up to 54 months).
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 0

17. Secondary Outcome: Primary Reason for Graft Loss
Description: The primary reason for graft loss was recorded by the Investigator. Graft loss was defined as graft failure (re-transplant) or participant death.
Time Frame: From enrollment until the end of study (up to 54 months).
Population: Participants in the modified full analysis set with graft loss.
Measure: Number; unit: participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 1
participants
  Recurrent disease | 0
  Death | 1

18. Secondary Outcome: Safety as Assessed by Clinical Signs and Symptoms, Laboratory Parameters and Diagnostic Tests
Description: An adverse event (AE) is defined as any reaction, side effect or other untoward medical occurrence, regardless of the relationship to study drug which occurred during the conduct of a clinical study. Clinically significant adverse changes in clinical status, routine laboratory studies or physical examinations were considered adverse events.
  A serious adverse event was any adverse event occurring at any dose that resulted in any of the following outcomes:
  * Death
  * Life-threatening adverse event
  * Inpatient hospitalization or prolongation of existing hospitalization
  * Persistent or significant disability or incapacity
  * Congenital abnormality or birth defect
  * Important medical event.
Time Frame: From the first dose of tacrolimus MR formulation through the last dose day plus 10 days (approximately 54 months).
Population: Modified safety analysis set defined as all participants who took at least 1 dose of both tacrolimus and tacrolimus MR formulation during the pharmacokinetic period of the study.
Measure: Number; unit: participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 18
participants
  Any adverse event | 12
  Any death | 1
  Any serious adverse event | 6
  Any AE leading to a change in study drug dose | 3
  AE leading to study drug discontinuation | 1

ADVERSE EVENTS:
Time Frame: From the first dose of tacrolimus MR through the last dose day plus 10 days (approximately 54 months).
Description: Adverse events are reported for the modified safety analysis set defined as all participants who took at least 1 dose of tacrolimus and one dose of tacrolimus MR during the pharmacokinetic period of the study.
Arm/Group | Tacrolimus MR
Serious Adverse Events (participants affected / at risk) | 6/18
Other Adverse Events (participants affected / at risk) | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus MR (N=18)
Bacteraemia (Infections and infestations) | 1
Pneumonia mycoplasmal (Infections and infestations) | 1
Pneumonia streptococcal (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Liver function test abnormal (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus MR (N=18)
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Tinea capitis (Infections and infestations) | 2
Viral upper respiratory tract infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Cat scratch disease (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Epstein-barr virus infection (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary tract infection staphylococcal (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Low density lipoprotein increased (Investigations) | 1
Weight increased (Investigations) | 1
Vomiting (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Pyrexia (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Glomerulosclerosis (Renal and urinary disorders) | 1
Maxillary sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Renal impairment (Renal and urinary disorders) | 1

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data or until 18 months have elapsed following study completion. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document.